CLINICAL TRIAL: NCT05540145
Title: Neo-Sequence 1: Phase 2 Study of Neoadjuvant Chemotherapy With or Without Antiangiogenesis and Sequential Immunotherapy for HER2-negative MMR-proficient Locally Advanced Gastric or Gastroesophageal Adenocarcinoma
Brief Title: Neo-Sequence 1: Neoadjuvant Chemotherapy With or Without Antiangiogenesis and Sequential Immunotherapy for HER2-negative MMR-proficient Locally Advanced Gastric or Gastroesophageal Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dong Bing Zhao, Clinical Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Other Study IDs: 21/489-3160
Record Dates: First submitted 2022-09-12; First posted 2022-09-14 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Gastric Cancer
Keywords: Neoadjuvant Chemotherapy; Immunotherapy; safety; Efficacy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood, fresh tumor tissue and fecal specimen at different time point;
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SOX plus Paclitaxel with or without antiangiogenesis followed by PD-1 antibody: SOX: Oxaliplatin+S-1
  Interventions: Drug: SOX plus Paclitaxel with or without antiangiogenesis followed by PD-1 antibody

INTERVENTIONS:
Drug: SOX plus Paclitaxel with or without antiangiogenesis followed by PD-1 antibody — Drug: Paclitaxel(albumin-bound) 130mg/m2, ivgtt, D1, Q2w Drug: Oxaliplatin 70 mg/m2, ivgtt, D1, q2w Drug: S-1 40mg (body surface area < 1.25m2), bid, D1-8, Q2w 50mg (body surface area >1.25m2, <1.5 m2), bid, D1-8, Q2w 60mg (body surface area >1.5m2), bid, D1-8, Q2w Drug: Bevacizumab, 5mg/kg, ivgtt, D1, Q14d Drug: PD-1 antibody, 200mg, ivgtt, D1, Q21d Patients with Her-2 negative, MMR-proficient locally advanced esophagogastric junction or gastric adenocarcinoma will receive 6 cycles of neoadjuvant chemotherapy with or without antiangiogenesis. After comprehensive evaluations, patients who respond to chemotherapy will further receive 2 cycles of PD-1 antibody comibed with antiangiogenesis and chemotherapy as neoadjuvant therapy.
  Drug: Pembrolizumab or sintilimab, 100~200mg, ivgtt, D1, Q3w. Patients will make the final decision of PD -1 antibody according to their economic condition.

SUMMARY:
This is a single-institution, prospective phase II trial designed to evaluate the efficacy of neoadjuvant chemotherapy and sequential immunotherapy in patients with locally advanced esophagogastric junction and gastric adenocarcinoma. Patients with Her-2 positive or dMMR tumors will be excluded from the study. Six cycles of nab-paclitaxel, oxaliplatin and S-1 with or without bevacizumab, followed by three circles of nab-paclitaxel, bevacizumab, with or without S-1 combined with two cycles of PD-1 monoclonal antibody, will be administered as neoadjuvant therapy. Patients will receive different adjuvant treatments depending on the degrees of surgical radicality and the pathological reactions of tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written (signed) informed consent;
2. Age ≥ 18 years and ≤75 years.
3. Has a pathologic diagnosis of gastroesophageal or gastric adenocarcinoma, mucinous adenocarcinoma or signet ring cell carcinoma.
4. Imaging (CT/ultrasonography of cervical lymph nodes and supraclavicular lymph nodes/ endoscopy and endoscopic ultrasound) confirmed at the stage of cT3/4a NanyM0(AJCC 8th).
5. Confirmed by immunohistochemistry (IHC) staining or genetic and transcriptional profiling detection to meet all of the following conditions:

   1. Her-2-negative was defined as IHC -, IHC 1+ or IHC 2+ and FISH negative;
   2. Mismatch repair-proficient (pMMR).
6. The Eastern Cooperative Oncology Group Performance status (ECOG PS) 0-1;
7. The main organ function meets the following criteria within 7 days before treatment:

   1. Hemoglobin (Hb) level ≥9.0 g/dl.
   2. Neutrophil count (ANC)≥1.5×10^9/L.
   3. Platelet (PLT) ≥100×10^9/L
   4. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) level ≤2.5×ULN.
   5. Serum creatinine (Cr) level ≤1.0×ULN and creatinine clearance ≥60 ml/min.
   6. Total bilirubin(TBIL) level ≤1.5×ULN.

Exclusion Criteria:

1. Confirmed at stage IV (AJCC 8th) or unresectable by investigator before enrolling.
2. Patienta have had prior chemotherapy, targeted small molecule therapy, or radiation therapy for the current diagnosis of EGJ cancer or gastric cancer.
3. Patients are allergic to study medication and its ingredients.
4. Patients have experienced or currently have other malignancies within 5 years.
5. Patients have an active infection requiring systemic therapy.
6. Women who are pregnant, breast-feeding or planning to become pregnant during treatment or within 6 months after treatment ends.
7. Patients have a history of psychotropic substance abuse and are unable to quit or have a mental disorder.
8. Patients with other severe acute or chronic conditions that may increase the risk of participation in the study and study treatment, or may interfere with interpretation of study results, and judged by the investigator as not suitable for participation in this clinical trial.
9. Diagnosis of immunodeficiency or active autoimmune disease, receiving or being treated with immunomodulators, systemic steroids or immunosuppressive drugs in the past two years.
10. Patients with gastrointestinal obstruction or uncontrolled bleeding undergo emergency surgery.
11. The proportion of other components in the pathology (such as squamous cell carcinoma, neuroendocrine carcinoma, etc.) exceeds 10%

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with endoscopically biopsy-proven Her-2(-), pMMR gastric cancer will receive preoperative neoadjuvant therapy.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Event-free survival (EFS) | From the recruitment to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
  The time from recruitment to any progression of disease precluding surgery, progression or recurrence of disease after surgery, progression of disease in the absence of surgery, or death from any cause.

SECONDARY OUTCOMES:
Major pathological response | From the date of recruitment to 3 months after all treatment ends
  It is defined as residual tumors less than 10% after neoadjuvant systemic therapy according to Mandard grade.
Overall survival(OS) | From the date of recruitment to the date of death from any cause or the date of last follow-up, assessed up to 36 months
  The time from recruitment to the date of death for any reason or the date of last follow-up
R0 resection rate | From the date of recruitment to 3 months after all treatment ends
  Rate of microscopically margin-negative resection
Adverse events | From the date of recruitment to 3 months after all treatment ends
  Adverse events (AEs) of neoadjuvant and adjuvant systemic therapy will be graded and documented according to NCI-CTCAE v5.0 and immune-related Adverse Event, irAE from the beginning of treatment to 3 months since the last dosage of treatment. Documentary will include severity, lasting period and occurrence time. Surgery complications will also be documented.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Beijing, Beijing Municipality, China